CLINICAL TRIAL: NCT02184455
Title: A Feasibility Study of DermGEN Dermal Regeneration Scaffold for the Treatment of Diabetic Foot Ulcers
Brief Title: Feasibility Study of DermGEN for Diabetic Foot Ulcer Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Paul F. Gratzer (Industry)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Dr. Paul F. Gratzer, CEO, DeCell Technologies Inc.
Organization: DeCell Technologies Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DeCell-001
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Results first posted 2019-09-16 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Type I; Diabetes Type II
Keywords: Diabetic; Chronic Ulcer; Wound Healing; Leg
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Diabetic type I/II patients with chronic ulcer present
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DermGEN Decellularized Dermal Matrix (Experimental): DermGEN is a product created by a patented process that decellularizes and sterilizes donated human tissue.
  Interventions: Biological: DermGEN

INTERVENTIONS:
Biological: DermGEN — DermGEN is a product created by a patented process that decellularizes and sterilizes donated human tissue.

SUMMARY:
The purpose of this clinical trial is to perform a limited pilot study to determine the safety and feasibility of DermGEN in the treatment of non-healing diabetic foot ulcers (DFU). This will be a one-arm prospective study. It is hypothesized that DermGEN treatment will result in positive healing outcomes with no significant adverse effects.

DETAILED DESCRIPTION:
This will be a one-arm prospective study. This study in Halifax will be mirrored in one other participating health care center in Toronto, Ontario, Canada with each centre anticipated to enrol 5-10 patients for a total of 15-20 patients.

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered eligible to participate in this study if each of the following inclusion criteria is satisfied:

1. Patient with documented stable Type I or II diabetes (HbA1C >7.0 within 1 month prior to Day 0).
2. Patient's ulcer has been present for a minimum of 2 weeks as of Day 0.
3. Study ulcer has healed <30% in size during the 2 weeks prior to Day 0.
4. Ulcer area is ≥1 cm2 prior to debridement at Day 0 of study.
5. Ulcer extends through dermis and into subcutaneous tissue but without exposure of muscle, tendon, bone or joint capsule.
6. Ulcer is free of necrotic debris and clinical infection, and is comprised of healthy vascular tissue suitable for skin grafting on Day 0.
7. Patient has adequate circulation to the foot as evidenced by palpable pulse or pulse detectable with Doppler ultrasound, and lack of visible cyanosis in skin bordering the ulcer.
8. Female patients are not pregnant at time of, or during study.
9. Patient and caregiver ready and willing to participate and comply with follow-up regime.
10. Patient or legal representative has read and signed the Institutional Ethics Review Board approved informed consent form.

Exclusion Criteria:

A subject will not be considered eligible to participate in this study if any one of the following exclusion criteria is satisfied:

1. Evidence of gangrene on affected foot.
2. Ulcer is over Charcot deformity (fractures or dislocation).
3. Ulcer is non-diabetic in etiology.
4. Ulcer has tunnels or sinus tracts that cannot be completely debrided.
5. Medical condition(s) that in the Investigator's opinion make the patient inappropriate for study
6. Patient has/had malignant disease not in remission for 5 years or more
7. Patient has acute or chronic hepatitis, cirrhosis, serum albumin <2.0 gm/dL, or has alkaline phosphatase or LDH at twice the normal upper limit
8. Patient receiving oral or parenteral corticosteroids, immunosuppression or cytotoxic agents, or is anticipated to require such agents during study
9. Patient received radiation therapy within 30 days of Day 0 of study
10. Patient has AIDS or is infected with HIV
11. Patient has participated in another study using investigational drug(s) or device within the previous 30 days
12. Obvious clinical signs and symptoms of ongoing cellulitis or osteomyelitis
13. Patient has any other condition which seriously compromises their ability to complete the study
14. Patient has known allergies to antibiotics, such as penicillin and streptomycin
15. Patient has a history of bleeding disorder
16. Patient received elective osseous procedures to the study foot within 30 days prior to screening visit, except that patients whose DFU overlies an area of treated osteomyelitis may be included, providing there exists a suitable base for application of the DermGEN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Glazebrook, PhD,MD, Principal Investigator — Queen Elizabeth II Health Sciences Center
Locations (2):
- Canada (2):
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Multi-disciplinary Leg Ulcer Clinic at the Queen Elizabeth II Hospital, Halifax, N.S. and Wound Care Clinic at St. Michael's Hospital, Toronto, O.N. The study was initiated on July 1st, 2016 and ended patient enrolment on March 31st, 2017.
Period: Overall Study
Arm/Group | DermGEN Decellularized Dermal Matrix
Started | 11
Completed | 10
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Baseline population was the same as intervention population
Arm/Group | DermGEN Decellularized Dermal Matrix
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Wound Area Reduction Compared to Baseline
Description: Digital photography was utilized to capture the appearance and size of the ulcer at each visit. In the photograph a measurement scale was shown beside the wound. The area of the wound was calculated by manually outlining wound edges on a digital image and then using the open source program ImageJ to calculate the area of the wound. For calculating the percentage change in area of the wound, the wound areas at each time point were divided by the size of the wound at baseline and multiplied by 100.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: percentage of wound closure
Arm/Group | DermGEN Decellularized Dermal Matrix
Number analyzed (Participants) | 10
percentage of wound closure | 87 (18)

2. Secondary Outcome: Percentage of Patients With Complete Healing at Any Time Point
Description: Complete healing is defined as 100% epithelialization without drainage. Digital photography was utilized to capture the appearance and size of the ulcer at each visit. In the photograph a measurement scale was shown beside the wound. The area of the wound was calculated by manually outlining wound edges on a digital image and then using the open source program ImageJ to calculate the area of the wound. For calculating the percentage change in area of the wound, the wound areas at each time point were divided by the size of the wound at baseline and multiplied by 100.
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DermGEN Decellularized Dermal Matrix
Number analyzed (Participants) | 10
Participants | 9

3. Secondary Outcome: Number of Patients With Adverse Events
Description: Reporting the number of patients participating in the study having adverse events
Time Frame: 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | DermGEN Decellularized Dermal Matrix
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Number of Patients With Ulcer Reoccurrence in the Same Location After Complete Healing
Description: Number of patients that reported a reoccurrence of the ulcer in the same location after complete healing at 1 year post treatment.
Time Frame: 1 year
Population: These are the number of patients that had their ulcer healed within the 20 weeks of the study.
Measure: Number; unit: participants
Arm/Group | DermGEN Decellularized Dermal Matrix
Number analyzed (Participants) | 9
participants | 9

5. Secondary Outcome: Percent Change in Wound Size Compared to Baseline
Description: Digital photography was utilized to capture the appearance and size of the ulcer at each visit. In the photograph a measurement scale was shown beside the wound. The area of the wound was calculated by manually outlining wound edges on a digital image and then using the open source program ImageJ to calculate the area of the wound. For calculating the percentage change in area of the wound, the wound areas at each time point were divided by the size of the wound at baseline and multiplied by 100. Note 100% equals complete closure of the wound.
Time Frame: 20 weeks
Measure: Mean (Standard Error); unit: percentage from baseline
Arm/Group | DermGEN Decellularized Dermal Matrix
Number analyzed (Participants) | 10
percentage from baseline | 92 (22)

6. Secondary Outcome: Percent Change in Wound Area From Baseline
Description: change in area of wound in percent from initial presentation
Time Frame: 12 Weeks
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | DermGEN Decellularized Dermal Matrix
Number analyzed (Participants) | 10
percentage of change from baseline | 97 (9)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the study and for up to 1 year post-treatment for all patients.
Arm/Group | DermGEN Decellularized Dermal Matrix
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
This study was a low numbered, one-arm, safety and feasibility study. No statistical analyses for superiority were intended nor attempted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT02184455/Prot_ICF_000.pdf